CLINICAL TRIAL: NCT04112225
Title: Testing the Effectiveness of an Online Behavioral Intervention in Reducing Loneliness
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Happify Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: None | Purpose: Other
Other Study IDs: 16
Record Dates: First submitted 2019-09-30; First posted 2019-10-02 (Actual); Last update posted 2020-09-02 (Actual); Status verified 2020-08

CONDITIONS: Psychological Distress; Loneliness

STUDY DESIGN:
Intervention Model Description: Users are randomly assigned between arms after completing baseline assessment and stay in that arm for the duration of the study.
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Positive affect condition (Active Comparator): Participants use Happify as it is currently available to consumers on the main site, including all engagement elements. Users may access a wide variety of 4-week programs and use them in any way they desire for the entire study period.
  Interventions: Behavioral: Happify
- Psychoeducation condition (Sham Comparator): Participants complete a series of quizzes and polls on Happify designed to engage them in thinking about well-being topics, but without giving any specific instructions for how to promote well-being. Participants gain access to 8 weeks worth of content, but may repeat the content as often as they like in the follow-up period.
  Interventions: Behavioral: Happify

INTERVENTIONS:
Behavioral: Happify — An online platform for conveying techniques from positive psychology, cognitive-behavioral therapy, and mindfulness-based stress reduction.

SUMMARY:
This study will use a longitudinal randomized experimental design. Participants will be randomly assigned to either a positive affect skills intervention or a psychoeducation control group and assessed with questionnaires at baseline and immediately post 8-week intervention.

DETAILED DESCRIPTION:
Participants will be randomly assigned to either a positive affect skills intervention or a psychoeducation control group, with each intervention lasting 8-weeks. Participants in the positive affect skills intervention will have full access to the unchanged Happify platform.

The psychoeducation control group participants will use a version of the Happify platform that encourages thinking about well-being through quizzes and polls without providing any instructions for promotion (i.e., Wait-list Control). Participants will be asked to complete questionnaires before and after the 8-week program, at which point study participation will end.

ELIGIBILITY:
Inclusion Criteria:

* No prior experience on the Happify platform (new user registration)
* Located in the United States
* Self reported loneliness/desire to be more connected to others

Exclusion Criteria:

* Participants who are under the age of 18, reside outside of the United States, have previously registered for Happify, or did not self report loneliness/desire to be more connected with others

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 890 (Actual)
Dates: Start 2019-08-01 (Actual); Primary Completion 2020-03-25 (Actual); Study Completion 2020-03-25 (Actual)

PRIMARY OUTCOMES:
Loneliness (Revised UCLA Loneliness Scale; Russell, Peplau, & Cutrona, 1980) | From start of 8-week intervention (baseline) to immediately post-intervention
  A 20-item scale designed to measure one's subjective feelings of loneliness as well as feelings of social isolation.

SECONDARY OUTCOMES:
Depression Patient Health Questionnaire (PHQ-9; Kroenke, Spitzer, & Williams, 2001) | From start of 8-week intervention (baseline) to immediately post-intervention
  A 9-item measure of depressive symptoms
Generalized Anxiety Disorder Screener (GAD-7; Spitzer, Kroenke, Williams, & Löwe, 2006) | From start of 8-week intervention (baseline) to immediately post-intervention
  A 7-item measure of anxiety symptoms
Perceived Stress Scale (PSS: Cohen, Kamarck, & Mermelstein, 1983) | From start of 8-week intervention (baseline) to immediately post-intervention
  10-item measure of perceived stress
Resilience(composite of Perceived Stress Scale [Cohen et al., 1983], Happify Scale [Carpenter et al., 2016] and Life Orientation Scale, Revised [Scheier & Carver, 1985]) | From start of 8-week intervention (baseline) to immediately post-intervention
  Composite score made of perceived stress, positive emotionality, and optimism. Perceived stress was measured using the Perceived Stress Scale (PSS; Cohen, Kamarck, & Mermelstein, 1983), a 10-item questionnaire that asks users to rate on a scale of 0 (never) to 4 (very often) how frequently they experience various symptoms of feeling stress. Positive emotionality was measured using the emotion subscale of the Happify Scale (HS-E; Carpenter, Crutchley, Zilca, Schwartz, Smith, Cobb, & Parks, 2016), which is a 4-item scale asking participants to rate the extent to which, over the past week, they have experienced positive and negative emotions that are activated or de-activated. Optimism was measured using the Life Orientation Scale, Revised (LOT-R; Scheier & Carver, 1985), a 6-item scale on which participants rate the extent to which they identify with optimistic or pessimistic beliefs.

CONTACTS AND LOCATIONS:
Overall Officials: Acacia Parks, PhD, Principal Investigator — Happify Inc.
Locations (1):
- Happify (an online platform -- study is entirely online), New York, New York, United States

IPD SHARING:
Plan to Share IPD: Undecided